CLINICAL TRIAL: NCT02685826
Title: A Phase 1/2 Multicenter, Open-label Study to Determine the Recommended Dose and Regimen of Durvalumab (MEDI4736) in Combination With Lenalidomide (LEN) With and Without Dexamethasone (DEX)in Subjects With Newly Diagnosed Multiple Myeloma (NDMM)
Brief Title: A Study of Durvalumab in Combination With Lenalidomide With and Without Dexamethasone in Adults With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDI4736-MM-002; 2015-004831-11 (EudraCT Number); U1111-1179-8722 (Registry Identifier: WHO)
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
Keywords: Open-label; Phase 1/2; Durvalumab; MEDI4736; Lenalidomide (Len); Dexamethasone (dex); Multiple Myeloma; Newly-Diagnosed (NDMM); Transplant Non-eligible (TNE); PD-L1; Durvalumab (DURVA)
MeSH Terms: conditions — Multiple Myeloma | interventions — durvalumab; Lenalidomide; Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A: High risk, TNE (Experimental): High risk, transplant non-eligible [TNE], newly diagnosed multiple myeloma (NDMM) participants who were administered
  * Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle
  * Oral lenalidomide (LEN) 25 mg/day (adjust per the creatinine clearance [CrCl]) value on Days 1 to 21 of each 28-day treatment cycle
  * Oral dexamethasone (dex) 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15, and 22 of each 28-day cycle
  Interventions: Drug: Durvalumab; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort B: >=65 years old, TNE (Experimental): >= 65 years old, transplant non-eligible [TNE], newly diagnosed multiple myeloma (NDMM) participants who were not high risk were administered
  * Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle
  * Oral lenalidomide (LEN) 25 mg/day (adjust per the creatinine clearance [CrCl]) value on Days 1 to 21 of each 28-day treatment cycle
  * Oral dexamethasone (dex) 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15, and 22 of each 28-day cycle, up to 12 cycles
  Interventions: Drug: Durvalumab; Drug: Lenalidomide; Drug: Dexamethasone
- Cohort C: High risk, Post-transplant (Experimental): High risk, post-transplant NDMM participants were administered the following as maintenance therapy:
  * Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle
  * Oral lenalidomide (LEN) 10 mg/day on Days 1 to 21 of each 28-day treatment cycle
  Interventions: Drug: Durvalumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Durvalumab — single use vials administered via intravenous infusion
  Other Names: MEDI4736; DUR, DURVA
Drug: Lenalidomide — capsules for oral administration
  Other Names: LEN; Revlimid
Drug: Dexamethasone — tablets for oral administration
  Other Names: corticosteroid; dex
  Arms: Cohort A: High risk, TNE; Cohort B: >=65 years old, TNE

SUMMARY:
This is a multicenter, open-label, Phase 1/2 study to determine the recommended dose and regimen of durvalumab in combination with lenalidomide (LEN) with and without dexamethasone (dex) in adults with newly diagnosed multiple myeloma (NDMM).

The study will consist of a dose-finding phase as well as a parallel dose-expansion phase to determine the optimal regimen.

******************************************************************************

The study was placed on full clinical hold by the United States (US) Food and Drug Administration (FDA) on 05 Sep 2017. The decision by the FDA was based on data from non-Celgene-sponsored studies related to risks of anti-programmed cell death 1 (PD-1), pembrolizumab, in combination with immunomodulatory agents. As the result, the study was closed for further enrollment, and all subjects were discontinued from all study treatments (durvalumab, lenalidomide and dexamethasone). All subjects are being followed for second primary malignancies (SPMs), every 6 months for 5 years after the last subject has been enrolled as per protocol. After stopping data collection in the clinical database, any SPM events will continue to be recorded in the subject's source documents, and reported to Celgene Drug Safety.

DETAILED DESCRIPTION:
The dose-finding phase will determine recommended dose (RD) for durvalumab in combination with lenalidomide (LEN) with and without dexamethasone (dex) in a 28-day treatment cycle. Three treatment Cohorts (A, B, and C) will be enrolled in parallel:

* Cohort A: durvalumab + LEN + dex in high risk transplant non-eligible (TNE) newly diagnosed multiple myeloma (NDMM) participants;
* Cohort B: durvalumab + LEN + dex (dex for up to 12 cycles) in ≥ 65 years old TNE NDMM participants who are not high risk;
* Cohort C: durvalumab + LEN as maintenance in post-transplant high risk NDMM participants.

Based on experience with durvalumab for other indications, the initial dose of durvalumab will be 1500 mg for each treatment cohort. The dose of durvalumab might be de-escalated to 750 mg level.

The dose of LEN will be 25 mg (adjustable per the creatinine clearance [CrCl] value) on Days 1 to 21 of each 28-day treatment cycle for participants in Cohort A and B. The dose of LEN will be 10 mg on Days 1 to 21 of each 28-day treatment cycle for participants in Cohort C.

The dose of dex will be 40 mg/day (for participants ≤ 75 years old) or 20 mg/day (for participants > 75 years old) on Days 1, 8, 15, and 22 of a 28-day cycle for Cohort A and Cohort B (for up to 12 cycles).

Initially, 6 participants will be enrolled into each cohort and each will receive 1500 mg durvalumab.

The dose-limiting toxicity (DLT) evaluation period will be the first treatment cycle.

* If ≤ 1 of the 6 initial participants experience a DLT within the first cycle, then the dose expansion phase may be initiated with durvalumab 1500 mg as the recommended dose (RD);
* If 2 or more of the 6 initial participants experience a DLT within the first cycle, then the maximum tolerated dose (MTD) has been exceeded and de-escalation to durvalumab 750 mg level after review of safety and pharmacokinetic/pharmacodynamic (PK/Pd) of the initial 6 participants by the Dose Review Team (DRT).

Any of the cohorts may be removed from the study based on emerging PK, Pd, efficacy or safety data.

Dose de-escalation will only occur after review of safety (DLT) and possibly PK/Pd data by the Dose Review Team ( DRT).

Note: In the US, two treatment arms (A and B) will be enrolled in parallel. Cohort C will enroll upon completion of at least 4 cycles of follow-up for safety assessment of Cohorts A and B.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled into the study:

  1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF)
  2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
  3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements
  4. Subject must have documented diagnosis with previously untreated (for cohort C, the induction and consolidation treatment along with the first autologous stem cell transplantation (ASCT) are allowed), symptomatic multiple myeloma (MM) as defined by the criteria below:

MM diagnostic criteria (all 3 required);

- Monoclonal protein present in the serum and/or urine

* Clonal bone marrow plasma cells ≥10% or biopsy-proven bony or extramedullary plasmacytoma
* Any one or more of the following myeloma defining events:

  1. one or more of the following Myeloma-related organ dysfunction (at least one of the following);
* (C) Calcium elevation (serum calcium >11.5 mg/dl )(>2.65 mmol/L)
* (R) Renal insufficiency (serum creatinine >2 mg/dl)(177 µmol/L or more) or creatinine clearance < 40 ml/min
* (A) Anemia (hemoglobin <10 g/dL or >2 g/dL below the lower limit of laboratory normal)
* (B) Bone lesions (lytic or osteopenic) one or more bone lesions on skeletal radiography, computed tomography (CT), or positron emission tomography-computed tomography (PET-CT)

  2. one or more of the following biomarkers of malignancy:
* Clonal bone marrow plasma cell percentage ≥60%
* Abnormal serum free light-chain ratio ≥100 (involved kappa) or < 0.01 (involved lambda)
* >1 focal lesions detected by functional imaging including PET/CT and/or whole body magnetic resonance imaging (MRI)

AND have measurable disease by protein electrophoresis analyses as defined by the following:

* Immunoglobulin G (IgG) MM: Serum monoclonal paraprotein (M-protein) level ≥ 1.0 g/dl or urine Mprotein level ≥ 200 mg/24 hours
* Immunoglobulin A (IgA) MM: Serum M-protein level ≥ 0.5 g/dl or urine M-protein level ≥ 200 mg/24 hours
* Immunoglobulin M (IgM) MM (IgM M-protein plus lytic bone disease documented by skeletal survey plain films): Serum M-protein level ≥ 1.0 g/dl or urine M-protein level ≥ 200 mg/24 hours
* Immunoglobulin D (IgD) MM: Serum M-protein level ≥ 0.05 g/dl or urine M-protein level ≥ 200 mg/24 hours
* Light chain MM: Serum M-protein level ≥ 1.0 g/dl or urine M-protein level ≥ 200 mg/24 hours

  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

  6. Females of childbearing potential (FCBP) must:

  a. Have two negative pregnancy tests as verified by the investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence from heterosexual contact.

  b. She must either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and be source documented) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study treatment, during the study therapy (including dose interruptions), and for 90 days after discontinuation of study treatment.

  c. Refrain from egg cell and blood donation for 90 days after the final dose of durvalumab.

  7. Male subjects must :

  a. Practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions and for at least 90 days following study treatment discontinuation, even if he has undergone a successful vasectomy.

  b. Refrain from sperm and blood donation for at least 90 days after the final dose of durvalumab.

  8. For Cohort A subject must be transplant non-eligible (TNE) and meet at least one of the following high risk factors:

  a. Cytogenetic abnormalities finding in malignant myeloma clone with t(4; 14); and / or del(17p); and / or 1q amplification; and / or t(14:16); or

  b. International Staging System (ISS) Stage III; or

  c. Serum lactate dehydrogenase (LDH) > 2*ULN (upper limit of normal).

  9. For Cohort B subject must be ≥ 65 years of age at the time of signing the informed consent form (ICF) and transplant non-eligible (TNE); excluding the subjects who meet the Cohort A criteria.

  10. For Cohort C subject must be after first autologous stem cell transplantation (ASCT) for NDMM and meet the following criteria:
  1. Have a post-transplant response as Partial response (PR) or better at the time of enrollment to this study;
  2. Have one of the following high risk factors at the time of NDMM diagnosis;
* Cytogenetic abnormalities finding in malignant myeloma clone with t(4; 14); and / or del(17p); and / or 1q amplification; and / or t(14; 16); or
* ISS stage III; or
* Serum LDH > 2*ULN;

  c. Minimal residual disease (MRD) positive (defined as more than 1 malignant cell in 105 cells) measured by ClonoSIGHT™NGS assay of a BMA sample) at the time of enrollment to this study; BMA sample collected at the time of multiple myeloma diagnosis, prior to induction therapy available for central MRD assessment by ClonoSIGHT™NGS assay

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid (ie, less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 14 days of Cycle 1 Day 1), for Cohort C, the induction and consolidation treatment along with the first Autologous stem cell transplantation (ASCT) are allowed)
  2. Any of the following laboratory abnormalities:

     1. Absolute neutrophil count (ANC) < 1,000/μL
     2. Untransfused platelet count < 75,000 cells/μL
     3. Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (SGOT/AST) or alanine aminotransferase (SGPT/ALT) > 2.5*upper limit of normal (ULN)
     4. Serum total bilirubin > 1.5*ULN or > 3.0 mg/dL for subjects with documented Gilbert's syndrome
     5. Corrected serum calcium >13.5 mg/dL (> 3.4 mmol/L)
  3. Renal failure requiring hemodialysis or peritoneal dialysis
  4. Any serious medical condition that places the subject at an unacceptable risk if he or she participates in this study. Examples of such a medical condition are, but are not limited to, subject with unstable cardiac disease as defined by: cardiac events such as myocardial infarction (MI) within the past 6 months, NYHA (New York Heart Association) heart failure class III-IV, uncontrolled atrial fibrillation or hypertension; subjects with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis and lupus, that likely need additional steroid or immunosuppressive treatments in addition to the study treatment
  5. Peripheral neuropathy ≥ Grade 2
  6. Primary AL (immunoglobulin light-chain) amyloidosis and myeloma complicated by amyloidosis
  7. Prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years with the exception of the following non-invasive malignancies:

     1. Basal cell carcinoma of the skin
     2. Squamous cell carcinoma of the skin
     3. Carcinoma in situ of the cervix
     4. Carcinoma in situ of the breast
     5. Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative
  8. Subjects is positive for human immunodeficiency virus (HIV); chronic or active hepatitis B or active hepatitis A, or C
  9. Subject had prior exposure to immunotherapy, including, but not limited to, other anti- CTLA-4,anti-PD-1, anti-PD-L1 monoclonal antibody or inhibitor, cell-based therapies, or cancer vaccines
  10. Subjects has history of organ or allogeneic stem cell transplantation
  11. Subjects who have had clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS multiple myeloma, or plasma cell leukemia
  12. Known or suspected hypersensitivity to the excipients contained in the formulation of durvalumab, lenalidomide, or dexamethasone
  13. Major surgery (as defined by the investigator) within the 28 days prior to the first dose of study treatment
  14. Received prior treatment (for any reason)with a monoclonal antibody within 5 half-lives of initiating study treatment
  15. Use of any investigational agents within 28 days or 5 half-lives (whichever is longer) of initiating study treatment
  16. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of study treatment. The following are exceptions to this criterion:

      1. Intranasal, inhaled, topical or local steroid injections (eg, intra-articular injection);
      2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent;
      3. Steroids as premedication for hypersensitivity reactions (eg, computed tomography (CT) scan premedication);
  17. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (eg, colitis, Crohn's disease], diverticulitis with the exception of a prior episode that has resolved or diverticulosis, celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener's syndrome [granulomatosis with polyangiitis); myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis, uveitis) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

      1. Subjects with vitiligo or alopecia;
      2. Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement; or
      3. Subjects with psoriasis not requiring systemic treatment;
  18. History of primary immunodeficiency
  19. Subject has incidence of gastrointestinal disease that may significantly alter the absorption of LEN
  20. Receipt of live, attenuated vaccine within 30 days prior to the first dose of durvalumab
  21. Unable or unwilling to undergo protocol required thromboembolism prophylaxis(for Cohort C, this will be only for the subjects who have a history of VTE)
  22. Females who are pregnant, nursing or breastfeeding, or intend to become pregnant during the participation to the study
  23. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
  24. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
  25. Any condition that confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (54):
- United States (7):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Carolinas Healthcare System, Charleston, South Carolina
  - Swedish Medical Center, Seattle, Washington
- Canada (9):
  - Local Institution - 206, Calgary, Alberta
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Local Institution - 203, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Local Institution - 202, Halifax, Nova Scotia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Local Institution - 205, Toronto, Ontario
  - Princess Margaret Hospital and University of Toronto, Toronto, Ontario
- Denmark (6):
  - Local Institution - 901, Copenhagen
  - Rigshospitalet University Hospital, Copenhagen
  - Local Institution - 903, Odense
  - Odense Universitetshospital, Odense
  - Local Institution - 902, Vejle
  - Vejle Hospital, Vejle
- Finland (2):
  - Helsinki UniversityCentral Hospital, Helsinki
  - Local Institution - 801, Helsinki
- Germany (5):
  - Universitatsklinikum Essen, Essen
  - Local Institution - 304, Koblenz
  - Praxis fuer Haematologie und Onkologie Koblenz, Koblenz
  - Local Institution - 302, Tübingen
  - University of Tubingen, Tübingen
- Italy (10):
  - Local Institution - 404, Rome, Roma
  - Local Institution - 405, Bologna
  - Policlinico S. Orsola, Bologna
  - I.R.C.C.S. Policlinico San Matteo - Universita di Pavia, Pavia
  - Local Institution - 402, Pavia
  - Local Institution - 403, Reggio Emilia
  - Servizio di Ematologia, A.O. - Arcispedale S.Maria Nuova, Reggio Emilia
  - Policlinico Agostino Gemelli, Rome
  - Azienda Ospedaliera San Giovanni Battista - Ospedale Molinette, Torino
  - Local Institution - 406, Torino
- Netherlands (4):
  - Local Institution - 704, Amsterdam
  - VU Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - Local Institution - 703, Rotterdam
- Spain (11):
  - Hopsital Germans Trias I Pujol, Badalona
  - Hospital 12 de Octobre, Madrid
  - Local Institution - 505, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Local Institution - 501, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Local Institution - 503, Salamanca
  - Hospital Doctor Peset, Valencia
  - Local Institution - 506, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Local Institution - 504, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: High Risk, TNE: High risk, transplant non-eligible [TNE], newly diagnosed multiple myeloma (NDMM) participants who were administered • Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle • Oral lenalidomide (LEN) 25 mg/day (adjust per the creatinine clearance [CrCl] value) on Days 1 to 21 of each 28-day treatment cycle • Oral dexamethasone (dex) 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15, and 22 of each 28-day cycle.
- Cohort B: >=65 Years Old, TNE: >= 65 years old, transplant non-eligible [TNE], newly diagnosed multiple myeloma (NDMM) participants who were not high risk were administered • Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle • Oral lenalidomide (LEN) 25 mg/day (adjust per the creatinine clearance [CrCl] value) on Days 1 to 21 of each 28-day treatment cycle • Oral dexamethasone (dex) 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15, and 22 of each 28-day cycle, up to 12 cycles.
- Cohort C: High Risk, Post-transplant: High risk, post-transplant NDMM participants were administered the following as maintenance therapy: • Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle • Oral lenalidomide (LEN) 10 mg/day on Days 1 to 21 of each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Started | 25 | 10 | 21
Completed (Completed treatment) | 0 | 0 | 0
Not Completed | 25 | 10 | 21
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Progressive Disease | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Full Clinical Hold by FDA | 19 | 9 | 20

BASELINE CHARACTERISTICS:
Population: Full analysis population. The Full Analysis Population (FAS) is defined as all participants who are enrolled (signed the inform consent form and meet all eligibility criteria) in the study. Participants are analyzed according to the initial cohort actually assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant | Total
Number analyzed (Participants) | 25 | 10 | 21 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (4.17) | 72.5 (5.25) | 59.6 (7.52) | 68.98 (9.33)
Age, Customized [Number; unit: participants]
  <=65 years | 0 | 0 | 17 | 17
  >65 years | 25 | 10 | 4 | 39
  <=75 years | 12 | 7 | 20 | 39
  >75 years | 13 | 3 | 1 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 0 | 4 | 19
  Male | 10 | 10 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 21 | 9 | 17 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 4 | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to assess how a subject's disease is progressing, and how the disease affects the daily living activities and determine appropriate treatment and prognosis. 0 = Fully Active, able to carry on all pre-disease performance without restriction; 1 = Restricted, in physically strenuous activity but ambulatory; 2 = Ambulatory and capable of all self-care; unable to carry out work activities; 3 = Capable of only limited self-care, confined to bed or chair >50% of waking hours; 4 = Completely Disabled, cannot carry on any self-care.
  Participants
    0 = Fully Active | 7 | 5 | 13 | 25
    1 = Restrictive but ambulatory | 14 | 5 | 8 | 27
    2 = ambulatory but unable to work | 4 | 0 | 0 | 4
International Staging System (ISS) for MM at Diagnosis [Count of Participants; unit: Participants] — Multiple myeloma has three stages, which are known as stage I, stage II and stage III. Staging in myeloma is done on the basis of the value of serum albumin and beta-2 microglobulin level. Stage I has the best prognosis and stage III the worst prognosis.
  Participants
    Stage I | 2 | 5 | 3 | 10
    Stage II | 7 | 5 | 7 | 19
    Stage III | 13 | 0 | 11 | 24
    Missing | 3 | 0 | 0 | 3
High-Risk Cytogenetic Abnormalities at Baseline [Count of Participants; unit: Participants]
  Yes | 17 | 0 | 2 | 19
  No | 8 | 10 | 19 | 37
Minimal Residual Disease (MRD) Status [Count of Participants; unit: Participants] — MRD status is either positive or negative. Positive was defined as more than 1 malignant cells in 10^5 cells as measured by the ClonoSIGHT(TM) NGS (next generation sequencing) assay of a bone marrow aspirate sample. Population: Data was collected for Cohort C only.
  Participants
    number analyzed (Participants) | 0 | 0 | 21 | 21
    Positive |  |  | 21 | 21
    Negative |  |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose-Limiting Toxicities (DLTs) During the Dose-Determining Timeframe (Day 1 - Day 28)
Description: A Dose Review Team (DRT) evaluated DLTs to determine the recommended dose (RD) of Durvalumab to use in the Expansion Period. A DLT was defined as: a. Grade 4 neutropenia for >= 5 days. b. Grade 3 neutropenia associated with fever (≥ 38.5°C / 101.3°F) of any duration. c. Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding, or platelets transfusion. d. Grade 4 hematologic toxicity that does not resolve to baseline level <=72 hours. e. Grade 4 anemia, unexplained by underlying disease. f. Any nonhematologic toxicity Grade ≥ 3 except for alopecia and nausea. g. Treatment interruption >= 2 weeks due to AE. If ≤ 1 of the 6 initial participants in each cohort experience a DLT during cycle 1, the RD was Durvalumab 1500 mg; If >=2 of the 6 initial participants in any cohort experience a DLT during cycle 1, the maximum tolerated dose (MTD) was exceeded and the dose level of Durvalumab was de-escalated to 750 mg
Time Frame: First treatment cycle: Day 1 to Day 28
Population: Dose-Determining Population consists of all participants from the Safety Population of the Dose Determining Period who received at least one dose of Durvalumab. Cohort B's Dose-Determining Population was 7 participants as one was considered non-evaluable and was therefore replaced per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 6 | 7 | 6
Participants | 1 | 1 | 0

2. Secondary Outcome: Participants With Treatment Emergent Adverse Events (TEAE)
Description: An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. A TEAE includes AEs between the first dose date of either study drug and 90 days after the last dose of study drug. A serious AE is any AE occurring at any dose that: • Results in death; • Is life-threatening; • Requires or prolongs existing inpatient hospitalization; • Results in persistent or significant disability/incapacity; • Is a congenital anomaly/birth defect; • Constitutes an important medical event. The Investigator assessed the relationship of each AE to study drug and graded the severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03): - Grade 1 = Mild - Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention required) - Grade 3 = Severe (limitation in activity; medical intervention required) - Grade 4 = Life-threatening - Grade 5 = Death
Time Frame: Day 1 up to Week 84 (the longer of 90 days after discontinuing treatment with DURVA, or 28 days after the last dose of LEN or dex)
Population: Safety population. The Safety Population is defined as all enrolled subjects who receive at least 1 dose of the study medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 25 | 10 | 21
Participants
  >= 1 TEAE | 24 | 9 | 18
  >=1 treatment-related TEAE | 22 | 8 | 17
  >=1 related to DURVA | 16 | 4 | 15
  >=1 related to LEN | 22 | 8 | 15
  >=1 related to dex | 16 | 6 | NA — Dexamethasone not administered to Cohort C
  >=1 TEAE of severity grade 3 or 4 | 19 | 8 | 7
  >=1 severity 3/4, related to study drug | 13 | 8 | 6
  >=1 severity 3/4, related to DURVA | 7 | 4 | 4
  >=1 severity 3/4, related to LEN | 11 | 8 | 4
  >=1 severity 3/4, related to dex | 5 | 2 | NA — Dexamethasone not administered to Cohort C
  >=1 Grade 5 TEAE (Death) | 1 | 0 | 1
  >=1 Grade 5 TEAE related to study drug | 0 | 0 | 1
  >=1 Grade 5 TEAE related to DURVA | 0 | 0 | 1
  >=1 Grade 5 TEAE related to LEN | 0 | 0 | 0
  >=1 Grade 5 TEAE related to dex | 0 | 0 | NA — Dexamethasone not administered to Cohort C
  >=1 Serious TEAE | 12 | 6 | 4
  >=1 Serious TEAE related to study drug | 8 | 4 | 4
  >=1 Serious TEAE related to DURVA | 5 | 1 | 4
  >=1 Serious TEAE related to LEN | 6 | 3 | 2
  >=1 Serious TEAE related to dex | 5 | 1 | NA — Dexamethasone not administered to Cohort C
  >=1 TEAE leading to discontinuation of study drug | 3 | 0 | 1
  >= TEAE leading to discontinuation of DURVA | 2 | 0 | 1
  >= TEAE leading to discontinuation of LEN | 3 | 0 | 0
  >= TEAE leading to discontinuation of dex | 2 | 0 | NA — Dexamethasone not administered to Cohort C
  >=1 leading to delay/reduction/interruption drug | 14 | 7 | 6
  >=1 leading to dose delay of DURVA | 10 | 3 | 4
  >=1 leading to infusion interruption of DURVA | 0 | 0 | 1
  >=1 leading to dose reduction of LEN | 2 | 2 | 3
  >=1 leading to interruption of LEN | 13 | 5 | 5
  >=1 leading to dose reduction of dex | 1 | 3 | NA — Dexamethasone not administered to Cohort C
  >=1 leading to interruption of dex | 9 | 3 | NA — Dexamethasone not administered to Cohort C

3. Secondary Outcome: Overall Response Rate (ORR) for Cohorts A and B: Percentage of Participants Who Achieved a Partial Response or Better According to the International Myeloma Working Group (IMWG) Uniform Response Criteria
Description: Tumor response, including progressive disease, was assessed by the investigators and captured the best assessment of response during the treatment period. ORR was defined as partial response (PR) or better which includes PR, very good partial response (VGPR), complete response (CR), or stringent complete response (sCR). A PR required ≥ 50% reduction of serum M-Protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours. If present at baseline, a ≥ 50% reduction in the size of soft tissue plasmacytomas was also required. sCR required - a negative immunofixation of serum and urine and - disappearance of any soft tissue plasmacytomas and - ≤ 5% plasma cells in bone marrow and normal free light-chain (FLC) ratio and - absence of clonal plasma cells by immunohistochemistry or 2- to 4-color flow cytometry.
Time Frame: Day 1 of each cycle starting with Cycle 2 up to Cycle 17 plus one week for the end of treatment visit (Day 29 up to Week 73)
Population: Efficacy Evaluable Population which consisted of enrolled participants who received at least 1 dose of the study medications and had at least 1 evaluable postbaseline response assessment. See the Response Improvement Rate outcome for an efficacy measure for Cohort C.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 24 | 10 | 0
percentage of participants | 66.7 [51.6 to 79.5] | 50.0 [26.7 to 73.3] |

4. Secondary Outcome: Response Improvement Rate (RIR) for Cohort C: Percentage of Participants Achieving a Response Improved From Cycle 1 Day 1 as Assessed by the Investigators Using the International Myeloma Working Group (IMWG) Uniform Response Criteria
Description: Response Improvement Rate is defined as the percentage of participants who achieved a response from treatment as compared to the pre-autologous stem cell transplantation [ASCT] diseases measurement used as baseline for response assessment. IMWG response categories could be stable disease (SD), partial response (PR), very good partial response (VGPR), complete response (CR), or stringent complete response (sCR), as long as it represented an improvement compared to prior to transplant.
Time Frame: Baseline (Cycle 1 Day 1); Treatment: Day 1 of each cycle starting with Cycle 2 up to Cycle 15 plus one week for the end of treatment visit (Day 29 up to Week 61)
Population: Efficacy Evaluable Population which consists of all enrolled participants who received at least 1 dose of the study medications and had at least 1 evaluable postbaseline response assessment.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 0 | 0 | 21
percentage of participants |  |  | 0 [NA to NA] — not estimable for a value of zero

5. Secondary Outcome: Time to Response (for Cohorts A and B)
Description: Time to response (for responders only, per IMWG Uniform Response Criteria) is calculated as the time from the first date of dosing of study medication to the first date of documented response (PR or better).
Time Frame: as for outcome 3
Population: Efficacy Evaluable Population: Participants in Cohorts A + B who had a response
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 16 | 5 | 0
weeks | 4.20 [3.9 to 23.1] | 4.10 [4.0 to 13.0] |

6. Secondary Outcome: Kaplan-Meier Estimates for Duration of Response (for Cohort A and B)
Description: Duration of response (for responders only) was defined as the time from earliest date of documented response (PR or better) to the earliest date of disease progression (DP) as determined by the investigator per IMWG Uniform Response criteria or death during study treatment, whichever occurred first.
Time Frame: as for outcome 3
Population: Efficacy Evaluable Population: Participants in Cohorts A + B who had a response.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 16 | 5 | 0
months | 10.3 [7.2 to NA] — not estimable since few responders had DP by the time the study was terminated | NA [NA to NA] — not estimable since no responder had DP by the time the study was terminated |

7. Secondary Outcome: Durvalumab (DURVA) Serum Pharmacokinetic (PK) Parameters in Cycle 1: Area Under the Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-last)
Description: Geometric mean was obtained by computing the arithmetic mean of the logarithm-transformed values of concentration/PK parameters and then using the exponentiation to return the computation to the original scales. Geometric CV% was calculated as follows: CV% = 100*SQRT(EXP(σ2)-1), where σ2 denotes the variance of the log-transformed values.
Time Frame: pre-infusion (-60 to -5 minutes prior to dose), end of infusion (EOI), 4 hours, 168 hours (Day 8), 336 hours (Day 15) and 504 hours (Day 22) after administration of DURVA on Day 1
Population: The PK Population included participants who received >=1 dose of study treatment and had >=1 measurable PK assessment. If participants were noncompliant with respect to dosing, had incomplete data, or other circumstances that would affect PK evaluation, inclusion was made on a case-by-case basis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/L
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 23 | 10 | 20
day*µg/L | 3535033.014 (39.8) | 3582905.960 (21.0) | 4026520.655 (39.1)

8. Secondary Outcome: Durvalumab (DURVA) Serum PK Parameters in Cycle 1: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/L
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 23 | 9 | 19
day*µg/L | 4944601.671 (60.9) | 5532568.144 (62.5) | 6531541.670 (36.4)

9. Secondary Outcome: Durvalumab (DURVA) Serum PK Parameters in Cycle 1: Maximum Observed Concentration (Cmax)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 23 | 10 | 20
µg/L | 449280.231 (36.7) | 452827.419 (25.5) | 482602.748 (39.9)

10. Secondary Outcome: Durvalumab (DURVA) Serum PK Parameters in Cycle 1: Time to Maximum Observed Concentration (Tmax)
Description: Time to maximum observed concentration of Durvalumab (DURVA) after multiple doses on day 1 obtained from the observed concentration versus time data
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: day
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 23 | 10 | 20
day | 0.051 [0.04 to 0.22] | 0.106 [0.04 to 0.22] | 0.180 [0.04 to 0.22]

11. Secondary Outcome: Durvalumab (DURVA) Serum PK Parameters in Cycle 1: Terminal Elimination Half-life (t1/2)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 23 | 9 | 19
day | 10.984 (52.1) | 13.376 (90.9) | 15.844 (29.8)

12. Secondary Outcome: Durvalumab (DURVA) Serum PK Parameters in Cycle 1: Clearance (CL)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 23 | 9 | 19
L/day | 0.303 (60.9) | 0.271 (62.5) | 0.230 (36.4)

13. Secondary Outcome: Durvalumab (DURVA) Serum PK Parameters in Cycle 1: Volume of Distribution (Vz)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 23 | 9 | 19
liters | 4.244 (33.5) | 4.582 (33.3) | 4.563 (42.9)

14. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 1: Area Under the Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-last)
Description: as for outcome 7
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 24 | 10 | 21
hour*ng/mL | 1468.102 (78.6) | 1442.549 (29.9) | 591.085 (22.3)

15. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 1: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf)
Description: as for outcome 7
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 13 | 3 | 12
hour*ng/mL | 2534.684 (48.6) | 2011.889 (26.8) | 768.104 (33.5)

16. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 1: Maximum Observed Concentration (Cmax)
Description: as for outcome 7
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 24 | 10 | 21
ng/mL | 395.774 (56.2) | 354.018 (34.7) | 161.372 (33.9)

17. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 1: Time to Maximum Observed Concentration (Tmax)
Description: Time to maximum observed concentration of Lenalidomide (LEN) after multiple doses on day 1 obtained from the observed concentration versus time data
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 24 | 10 | 21
hour | 1.050 [0.42 to 4.08] | 1.925 [0.50 to 4.00] | 1.150 [0.43 to 4.17]

18. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 1: Terminal Elimination Half-life (t1/2)
Description: as for outcome 7
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 13 | 3 | 12
hour | 3.477 (61.3) | 3.051 (16.8) | 2.883 (29.2)

19. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 1: Apparent Clearance (CL/F)
Description: as for outcome 7
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 13 | 3 | 12
L/hour | 8.838 (52.7) | 12.426 (26.8) | 13.019 (33.5)

20. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 1: Apparent Volume of Distribution (Vz/F)
Description: as for outcome 7
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 13 | 3 | 12
liters | 44.329 (25.4) | 54.689 (29.7) | 54.157 (22.3)

21. Secondary Outcome: Lenalidomide (LEN) Plasma PK Parameters in Cycle 1 Day 15: Area Under the Concentration-time Curve From Time Zero to the Last Measured Time Point (AUC0-last)
Description: as for outcome 7
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 18 | 9 | 16
hour*ng/mL | 1911.739 (65.5) | 1754.349 (34.3) | 629.151 (16.8)

22. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 15: Maximum Observed Concentration (Cmax)
Description: as for outcome 7
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 18 | 9 | 16
ng/mL | 409.764 (66.0) | 452.850 (31.7) | 171.235 (33.6)

23. Secondary Outcome: Lenalidomide (LEN) Plasma Pharmacokinetic (PK) Parameters in Cycle 1 Day 15: Time to Maximum Observed Concentration (Tmax)
Description: Time to maximum observed concentration of Lenalidomide (LEN) after multiple doses on day 15 obtained from the observed concentration versus time data
Time Frame: Cycle 1 Day 15: pre-dose, 0.5, 1, 2, 4, and 8 hours post LEN dose
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 18 | 9 | 16
hour | 2.000 [1.00 to 8.00] | 1.000 [0.55 to 2.00] | 1.042 [0.47 to 4.00]

24. Secondary Outcome: Participants Who Developed Anti-drug Antibody Against Durvalumab
Description: The number of participants who develop antidrug antibody against durvalumab at any of the sampling timepoints during the study.
Time Frame: Pre-dose samples on Day 1 of cycles 1, 2, 4, 6, 10, and 14 (study days 1, 29, 85, 141, 253, 393)
Population: The Safety Population was defined as all enrolled participants who receive at least 1 dose of the study medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 25 | 10 | 21
Participants | 0 | 1 | 0

25. Secondary Outcome: Participants Who Had Either Disease Progression or Death
Description: This outcome was originally defined as a Kaplan-Meier estimate of progression-free survival (PFS) which estimated the time between first date of dosing of study medication and disease progression, as determined by the investigator using the IMWG Uniform Response Criteria, or death during study treatment, whichever occurred earlier. However due to the early study termination and limited follow-up time, the majority of participants were censored for PFS analysis. Data reported instead represent the number of participants who died during study treatment or had disease progression within 90 days of the last dose of durvalumab.
Time Frame: Day 1 up to Week 84
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 25 | 10 | 21
Participants | 4 | 1 | 3

26. Secondary Outcome: Participants Who Died Up To Data Cut-off Date (15 December 2017)
Description: This outcome was originally defined as a Kaplan-Meier estimate of overall survival (OS) and was defined as the time between first date of dosing of study medication and death due to any cause. However due to the early study termination and limited follow-up time, the majority of participants were censored for OS analysis. Data reported instead represent the number of participants who died due to any cause from Day 1 up to data cut-off.
Time Frame: Day 1 up to Week 87
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
Number analyzed (Participants) | 25 | 10 | 21
Participants | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs are assessed from first dose up to week 84 (the longer of 90 days after discontinuing treatment with DURVA, or 28 days after the last dose of LEN or DEX). Participants were assessed for all-cause mortality from their first dose to their study completion (Up to approximately 88 months).
Groups:
- Cohort A: High Risk, TNE: High risk, transplant non-eligible [TNE], newly diagnosed multiple myeloma (NDMM) participants who were administered - Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle - Oral lenalidomide (LEN) 25 mg/day (adjust per the creatinine clearance [CrCl] value) on Days 1 to 21 of each 28-day treatment cycle - Oral dexamethasone (dex) 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15, and 22 of each 28-day cycle.
- Cohort B: >=65 Years Old, TNE: >= 65 years old, transplant non-eligible [TNE], newly diagnosed multiple myeloma (NDMM) participants who were not high risk were administered - Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle - Oral lenalidomide (LEN) 25 mg/day (adjust per the creatinine clearance [CrCl] value) on Days 1 to 21 of each 28-day treatment cycle - Oral dexamethasone (dex) 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15, and 22 of each 28-day cycle, up to 12 cycles.
- Cohort C: High Risk, Post-transplant: High risk, post-transplant NDMM participants were administered the following as maintenance therapy: Intravenous (IV) durvalumab at 1500 mg on Day 1 of each 28-day cycle Oral lenalidomide (LEN) 10 mg/day on Days 1 to 21 of each 28-day treatment cycle.
Arm/Group | Cohort A: High Risk, TNE | Cohort B: >=65 Years Old, TNE | Cohort C: High Risk, Post-transplant
All-Cause Mortality (participants affected / at risk) | 9/25 | 3/10 | 5/21
Serious Adverse Events (participants affected / at risk) | 12/25 | 6/10 | 4/21
Other Adverse Events (participants affected / at risk) | 24/25 | 9/10 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: High Risk, TNE (N=25) | Cohort B: >=65 Years Old, TNE (N=10) | Cohort C: High Risk, Post-transplant (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Cystitis klebsiella (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: High Risk, TNE (N=25) | Cohort B: >=65 Years Old, TNE (N=10) | Cohort C: High Risk, Post-transplant (N=21)
Anaemia (Blood and lymphatic system disorders) | 13 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 11 | 5 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 6
Hypothyroidism (Endocrine disorders) | 2 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 13 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 2 | 2
Asthenia (General disorders) | 7 | 2 | 1
Chills (General disorders) | 1 | 0 | 2
Fatigue (General disorders) | 4 | 3 | 7
General physical health deterioration (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 8 | 2 | 0
Peripheral swelling (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 3 | 4 | 3
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 5 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1
Amylase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 3 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 5 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 3
Dysgeusia (Nervous system disorders) | 3 | 1 | 2
Headache (Nervous system disorders) | 1 | 2 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 2
Tremor (Nervous system disorders) | 3 | 1 | 0
Depression (Psychiatric disorders) | 4 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 4 | 3
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was placed on full clinical hold by the United States (US) Food and Drug Administration (FDA) on 05 Sep 2017. As the result, the study was closed for further enrollment, and all participants were discontinued from all study treatments (durvalumab, lenalidomide and dexamethasone). All participants were followed for second primary malignancies (SPMs), every 6 months for 5 years after the last participant has been enrolled as per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02685826/Prot_002.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT02685826/SAP_001.pdf